CLINICAL TRIAL: NCT03425838
Title: BOOG 2017-03: Endocrine Therapy Plus CDK 4/6 Inhibition in First- or Second-line for Hormone Receptor Positive Advanced Breast Cancer - the SONIA Study
Brief Title: Endocrine Therapy Plus CDK4/6 in First or Second Line for Hormone (SONIA) Receptor Positive Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Borstkanker Onderzoek Groep (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2017-03; 2017-002334-23 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2018-02-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Female
Keywords: CDK 4/6 inhibitor
MeSH Terms: interventions — palbociclib; Letrozole; Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strategy A CDK4/6 inhibitor in 1st line (Active Comparator): Non-steroidal aromatase inhibitor (letrozole or anastrozole, at the discretion of the treating physician) plus CDK4/6 inhibitor (palbociclib, ribociclib or abemaciclib, depending on availability and physician's preference) in first line followed by fulvestrant in second line.
  Interventions: Drug: CDK 4/6 inhibitor; Drug: Non-Steroidal Aromatase Inhibitor; Drug: Fulvestrant
- Strategy B CDK4/6 inhibitor in 2nd line (Active Comparator): Non-steroidal aromatase inhibitor (letrozole or anastrozole, at the discretion of the treating physician) in first line followed by fulvestrant plus CDK4/6 inhibitor in second line (palbociclib, ribociclib or abemaciclib, depending on availability and physician's preference).
  Interventions: Drug: CDK 4/6 inhibitor; Drug: Non-Steroidal Aromatase Inhibitor; Drug: Fulvestrant

INTERVENTIONS:
Drug: CDK 4/6 inhibitor — Adding CDK 4/6 inhibitor (pabociclib, ribociclib or abemaciclib depending on availability and physician's preference) to either first line treatment (with non-steroidal aromatase inhibitors, either letrozole or anastrozole) or second line treatment (with fulvestrant) in advanced HR+/HER2-negative breast cancer
  Other Names: palbociclib,Ibrance,ribociclib,Kisqali,abemaciclib,Verzenio
Drug: Non-Steroidal Aromatase Inhibitor — Adding CDK 4/6 inhibitor (pabociclib, ribociclib or abemaciclib depending on availability and physician's preference) to either first line treatment (with non-steroidal aromatase inhibitors, either letrozole or anastrozole) or second line treatment (with fulvestrant) in advanced HR+/HER2-negative breast cancer
  Other Names: NSAI, letrozole, Femara®, anastrozole, Arimidex®
Drug: Fulvestrant — Adding CDK 4/6 inhibitor (pabociclib, ribociclib or abemaciclib depending on availability and physician's preference) to either first line treatment (with non-steroidal aromatase inhibitors, either letrozole or anastrozole) or second line treatment (with fulvestrant) in advanced HR+/HER2-negative breast cancer
  Other Names: SERD, Faslodex®

SUMMARY:
Given the uncertain benefit in efficacy of adding CDK 4/6 to first rather than second line endocrine treatment, the aim of this project is to evaluate whether the sequence of an aromatase inhibitor plus CDK 4/6 in first line followed by fulvestrant in second line is superior to the sequence of an aromatase inhibitor in first line followed by fulvestrant plus CDK4/6 in second line.

DETAILED DESCRIPTION:
Combining cyclin-dependent kinases 4 and 6 (CDK 4/6) inhibitors with endocrine therapies in hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative advanced breast cancer has shown to result in substantial improvements in progression-free survival. There is however no evidence that this combination strategy leads to an improved overall survival. Furthermore, no specific subgroups that will or will not benefit from the combination of drugs have been identified yet. This means the optimal strategy for deploying CDK 4/6 inhibitors in clinical practice is not yet known. Since CDK 4/6 inhibitors are costly and can have toxic effects, it is important to determine the optimal treatment strategy to avoid both over- and undertreatment.

The SONIA-trial is an investigator-initiated, multicenter, randomized phase III study. The primary objective of this study is to evaluate if treatment with a non-steroidal aromatase inhibitor combined with CDK 4/6 inhibition in first line followed at progression by fulvestrant in second line (strategy A) improves progression-free survival compared to treatment with a non-steroidal aromatase inhibitor in first line followed at progression by fulvestrant combined with CDK4/6 inhibition in second line (strategy B). The primary end point is progression-free survival after two lines (PFS2), secondary end points include overall survival, quality of life, safety and biomarker analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥ 18 years of age) with proven diagnosis of adenocarcinoma of the breast with evidence of loco-regional recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent and for whom chemotherapy is not clinically indicated.
2. Documentation of histologically or cytologically confirmed diagnosis of estrogen-receptor (ER) expression >10% and/or progesterone receptor (PR) expression >10% breast cancer based on local laboratory results.
3. Previously untreated with any systemic anti-cancer therapy for loco-regional recurrent or metastatic HR+ disease, with the exception of recently started (within 28 days of randomization) endocrine therapy.
4. Women who are not post-menopausal must use LHRH agonist. Postmenopausal status is defined as:

   1. prior bilateral surgical oophorectomy, or
   2. spontaneous cessation of regular menses for at least 12 consecutive months without OAC
   3. in case of doubt serum estradiol <20 umol/l and follicle stimulating hormone (FSH) levels >15 IU/L at screening
5. Measurable or evaluable disease as defined per RECIST v.1.1 (see Appendix 3) or bone-only disease. Tumor lesions previously irradiated or subjected to other locoregional therapy will only be deemed measurable if disease progression at the treated site after completion of therapy is clearly documented.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
7. Adequate organ and marrow function defined as follows:

   1. ANC ≥1,000/mm3 (1.0 x 10e9 /L);
   2. Platelets ≥50,000/mm3 (50 x 10e9 /L);
   3. Estimated creatinine clearance ≥ 30 mL/min as calculated using the method standard for the institution;
   4. Total serum bilirubin ≤1.5 x ULN (≤3.0 x ULN if Gilbert's disease);
   5. AST and ALT ≤3 x ULN (≤5.0 x ULN if liver metastases present);
8. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade ≤1, except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion.
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
10. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legal representative) has been informed of all pertinent aspects of the study before any study-specific activity is performed.

Exclusion Criteria:

1. Patients with advanced, symptomatic, visceral spread, who are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% liver involvement).
2. Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (e.g., radiotherapy, stereotactic surgery) and are clinically stable without the use of steroids for at least 4 weeks before randomization
3. Prior neoadjuvant or adjuvant treatment with an aromatase inhibitor (i.e., anastrozole, letrozole or exemestane) with disease recurrence while on or within 12 months of treatment.
4. Prior treatment with any CDK4/6 inhibitor.
5. Patients treated within the last 7 days prior to randomization with:

   1. Food or drugs that are known to be CYP3A4 inhibitors (ie, amprenavir, atazanavir, boceprevir, clarithromycin, conivaptan, delavirdine, diltiazem, erythromycin, fosamprenavir, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, verapamil, voriconazole, and grapefruit or grapefruit juice);
   2. Drugs that are known to be CYP3A4 inducers (ie, carbamazepine, felbamate, nevirapine, phenobarbital, phenytoin, primidone, rifabutin, rifampin, rifapentin, and St. John's wort).
6. Major surgery, chemotherapy, radiotherapy, any investigational agents, or other anti-cancer therapy within 2 weeks before randomization. Patients who received prior radiotherapy to ≥25% of bone marrow are not eligible independent of when it was received.
7. Diagnosis of any other malignancy prior to randomization, except those that are not believed to influence the patient's prognosis and do not require any further treatment. This includes, but is not limited to adequately treated basal cell or squamous cell skin cancer and carcinoma in situ of the cervix.
8. QTc >480 msec at baseline
9. Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or any upper gastrointestinal surgery including gastric resection.
10. Known hypersensitivity to letrozole or anastrozole, or any of its excipients, or to any palbociclib excipients.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
12. Recent or active suicidal ideation or behavior.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PFS2 | Until objective disease progression, symptomatic deterioration, or unacceptable toxicity on second line treatment, death, strategy violation, or withdrawal of consent, whichever occurs first, assessed up to 60 months
  Progression-free survival after two lines of treatment (PFS2)

SECONDARY OUTCOMES:
OS | Date of randomization until date of death due to any cause, assessed up to 60 months
  Overall survival
FACT-B questionnaire | Questionnaires will be administered at baseline and thereafter every three months, up to 60 months
  Quality of Life questionnaire
EQ-5D questionnaire | Questionnaires will be administered at baseline and thereafter every three months, up to 60 months
  Quality of Life questionnaire
iMTA RUQ-B questionnaire | Questionnaires will be administered at baseline and thereafter every six months, up to 60 months
  Quality of Life questionnaire
Number of participants with grade 3 or 4 treatment-related neutropenia as assessed by CTCAE v4.0 | Through study completion, assessed up to 60 months
  Safety assessment will consist of monitoring of all grade 3 and grade 4 neutropenia (absolute neutrophil count/L)
Number of participants with grade 3 or 4 treatment-related thrombocytopenia as assessed by CTCAE v4.0 | Through study completion, assessed up to 60 months
  Safety assessment will consist of monitoring of all grade 3 and grade 4 thrombocytopenia (platelet count/L)
Number of participants with grade 3 or 4 treatment-related anemia as assessed by CTCAE v4.0 | Through study completion, assessed up to 60 months
  Safety assessment will consist of monitoring of all grade 3 and grade 4 anemia (mmol/L)
Number of participants with grade 3 or 4 treatment-related elevated liver enzymes (ALAT/ASAT/AF/GGT/bilirubin) as assessed by CTCAE v4.0 | Through study completion, assessed up to 60 months
  Safety assessment will consist of monitoring of all grade 3 and grade 4 elevated liver enzymes (elevation compared to upper limit of normal)
Number of participants with grade 3 or 4 treatment-related other toxicities as defined in CTCAE v4.0 | Through study completion, assessed up to 60 months
  Safety assessment will consist of monitoring of all grade 3 and grade 4 other toxicities as defined in CTCAE v4.0
Cost-effectiveness by means of a decision model (a multistate Markov model or a Discrete Event Simulation model) | At 60 months after entry into the study
  The cost and outcomes of both arms will be assessed by means of a decision model (a multistate Markov model or a Discrete Event Simulation model). Cost-effectiveness will be determined by comparing costs and effects of both treatment strategies. Quality adjusted life years will be computed by multiplying life-years with the observed utility scores during those life years. The friction cost method will be used for estimating the societal costs of productivity losses. Unit costs for drugs will be derived from www.medicijnkosten.nl or the Z-index. The costs of a hospital day, outpatient visit, and day care treatment, will be based on the Dutch costing manual. Other costs will be collected from NZA tariffs. All costs will be expressed in Euros.
ORR | Through study completion, assessed up to 60 months
  Objective response rate
Plasma through levels | Through study completement
  Plasma through levels of CDK4/6 inhibitor measured in blood samples obtained at cycle 1, day 15 (of 28 days in one cycle) and at cycle 2, day 15 in participants treated with CDK4/6 inhibitors.
Pharmacogenomics | On day 15 of cycle 1 (a cycle is 28 days)
  DNA sequencing in a blood sample obtained at cycle 1, day 15 (of 28 days in one cycle) of treatment with CDK4/6 inhibitor.
Liquid biopsies | At baseline of first line, at cycle 1 day 15 (a cycle is 28 days), at cycle 4 day 1, at baseline of second line, at cycle 1 day 15 (a cycle is 28 days), at cycle 4 day 1 and at disease progression
  Circulating tumor DNA isolated from blood samples collected at 7 timepoints during the study. Mutation level during the study and at disease progression will be compared to base-line mutation level.
Tissue microarray | At baseline
  Tissue microarray on archived FFPE tissue blocks of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: A. Jager, MD, PhD, Principal Investigator — Borstkanker Onderzoek Groep; A E van Leeuwen-Stok, PhD, Study Director — BOOG Study Center
Locations (72):
- Netherlands (72):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwestziekenhuisgroep, Alkmaar
  - ZGT, Almelo
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - Nki - Avl, Amsterdam
  - VUmc, Amsterdam
  - AMC, Amsterdam
  - BovenIJ Ziekenhuis, Amsterdam
  - OLVG, Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Wilhelmina ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Alexander Monro Ziekenhuis, Bilthoven
  - Maasziekenhuis Pantein, Boxmeer
  - Amphia, Breda
  - IJsselland, Capelle aan den IJssel
  - Reinier de Graaf, Delft
  - Deventer Ziekenhuis, Deventer
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Nij Smellinghe, Drachten
  - Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Treant Zorggroep, Emmen
  - Medisch Spectrum Twente, Enschede
  - St. Anna Ziekenhuis, Geldrop
  - Admiraal de Ruyter, Goes
  - Rivas Beatrixziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - UMC Groningen, Groningen
  - Ropcke Zweers, Hardenberg
  - Sint Jansdal, Harderwijk
  - Tjongerschans, Heerenveen
  - Elkerliek ziekenhuis, Helmond
  - Tergooi, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Dijklander Ziekenhuis, Hoorn
  - MC Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, Leiden
  - LUMC, Leiden
  - St. Antonius, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Radboudumc, Nijmegen
  - Laurentius, Roermond
  - Bravis ziekenhuis, Roosendaal
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Ikazia, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Zuyderland, Sittard
  - Antonius Ziekenhuis, Sneek
  - Spijkenisse Medisch Centrum, Spijkenisse
  - ZorgSaam, Terneuzen
  - Haaglanden Medisch Centrum, The Hague
  - HaGaziekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth Tweesteden, Tilburg
  - Bernhoven, Uden
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht
  - VieCuri, Venlo
  - St. Jans Gasthuis, Weert
  - Streekziekenhuis Koningin Beatrix, Winterswijk
  - Zaans Medisch Centrum, Zaandam
  - Langeland, Zoetermeer
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Derived] Wortelboer N, Kent S, Blommestein HM, van Ommen-Nijhof A, van der Noort V, van den Pol E, Paez CG, Beeker A, Beelen K, Hamming LC, Heijns JB, Honkoop AH, de Jong PC, van Rossum-Schornagel QC, van de Mheen CVS, Tol J, Driel CST, Vrijaldenhoven S, van Leeuwen-Stok AE, Sonke GS, Jager A, Konings IR. Health-related quality of life with first- vs second-line CDK4/6 inhibitor use in advanced breast cancer: results from the SONIA trial. J Natl Cancer Inst. 2025 Nov 21:djaf334. doi: 10.1093/jnci/djaf334. Online ahead of print. PMID 41270788
- [Derived] Wortelboer N, Kent S, Konings IR, van Ommen-Nijhof A, van der Noort V, van den Pol E, Guerrero Paez C, van Bekkum ML, van den Berkmortel FWPJ, Droogendijk HJ, Houtsma D, Oosterkamp HM, van der Padt-Pruijsten A, Siemerink EJM, Tol J, van Zweeden AA, van Leeuwen-Stok AE, Sonke GS, Jager A, Blommestein HM. Health economic outcomes and costs of CDK4/6 inhibitor use in first- versus second-line for advanced breast cancer: A cost-effectiveness analysis of the phase 3 SONIA trial. Eur J Cancer. 2025 Dec 9;231:116051. doi: 10.1016/j.ejca.2025.116051. Epub 2025 Oct 25. PMID 41207182
- [Derived] Jongbloed EM, Wortelboer N, de Weerd V, Beaufort CM, Ruigrok-Ritstier K, Van MN, Kraan J, van Zweeden AA, van der Padt-Pruijsten A, Hamming LC, Konings IR, Sonke GS, Oomen-de Hoop E, Martens JWM, Jager A, Wilting SM. Early versus deferred use of CDK4/6 inhibitors in advanced breast cancer: circulating tumor DNA analysis of a randomized phase 3 trial. Nat Med. 2025 Nov;31(11):3662-3667. doi: 10.1038/s41591-025-03935-w. Epub 2025 Sep 4. PMID 40908356
- [Derived] van Ommen-Nijhof A, Konings IR, van Zeijl CJJ, Uyl-de Groot CA, van der Noort V, Jager A, Sonke GS; SONIA study steering committee. Selecting the optimal position of CDK4/6 inhibitors in hormone receptor-positive advanced breast cancer - the SONIA study: study protocol for a randomized controlled trial. BMC Cancer. 2018 Nov 20;18(1):1146. doi: 10.1186/s12885-018-4978-1. PMID 30458732